CLINICAL TRIAL: NCT02846935
Title: p53/p16-Independent Epigenetic Therapy With Oral Decitabine/Tetrahydrouridine for Refractory/Relapsed Lymphoid Malignancies
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yogen Saunthararajah (Other)
Responsible Party: Sponsor-Investigator, Yogen Saunthararajah, Professor of Hematology and Oncology, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1416
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: T-cell Lymphoma; Aggressive B-cell Lymphoma; Non-Hodgkin's Lymphomas; Indolent B-cell Lymphoma
Keywords: p16/CDKN2A; TP53; THU; Decitabine; Tetrahydrouridine; DEC
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — Decitabine; Tetrahydrouridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Decitabine + Tetrahydrouridine (Experimental): oral THU dosed by weight, followed by oral decitabine dosed by weight for 60 minutes (± 10 minutes) after the THU, twice weekly on consecutive days.
  Treatment on protocol monitoring continues for 52 weeks.
  Interventions: Drug: Decitabine; Drug: Tetrahydrouridine

INTERVENTIONS:
Drug: Decitabine — 2-4 capsules depending on the weight of participant. Dec capsules are ingested ~60 minutes after THU capsules.
  Other Names: DEC
Drug: Tetrahydrouridine — 2-4 capsules depending on the weight of participant. Oral THU capsules followed 60 minutes later by oral Dec capsules are ingested 2X/week on consecutive days.
  Other Names: THU

SUMMARY:
The purpose of this study is to evaluate how well the study drug works and safety of oral decitabine in patients with refractory or relapsed lymphoid malignancies. The decitabine is being given at a lower dose than used for its approved use. It is also being given with another drug, tetrahydrouridine (THU), to improve the exposure of lymphoma cells to decitabine.

DETAILED DESCRIPTION:
Primary objective: To determine the objective response rate to oral THU-Dec in patients with 3 separate biologic subsets of refractory/relapsed lymphoid malignancies:

1. T-cell lymphoma,
2. Aggressive B cell lymphoma,
3. indolent B-cell lymphoma .

Secondary objectives:

(i) To evaluate the toxicity of oral THU-Dec in these patients; (ii) To evaluate hypotheses regarding mechanisms of resistance and predictive biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-proven T- or B-cell lymphoma
* Subjects must have received 1 or more prior therapies for this disease and have had stable disease or progressive disease based upon the criteria from the Revised Response Criteria for Malignant Lymphoma78, or intolerable toxicities precluding further therapy with a prior regimen
* Subjects must have measurable disease per Revised Response Criteria for Malignant Lymphoma78
* ECOG performance status 0 - 2
* Adequate organ function as defined by the following criteria:

  * Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x laboratory upper limit of normal (ULN)
  * Total serum bilirubin ≤ 2.0 x ULN (except if Gilbert's disease)
  * Absolute neutrophil count (ANC) ≥ 1500/uL
  * Platelets ≥ 50,000/uL
  * Hemoglobin ≥ 8.0 g/dL (transfusion permitted)
  * Serum calcium ≤ 12.0 mg/dL
  * Serum Creatinine ≤ 3.0 mg/dL
* Patients with history of CNS lymphoma can be enrolled if the CNS disease has been controlled with therapy for a minimum of 4 weeks. Brain MRI is not required for eligibility.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Life expectancy ≤ 4 months in the judgment of the treating clinician
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness (HIV-positive subjects on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with oral THU-Dec. Appropriate studies will be undertaken in subjects receiving combination antiretroviral therapy when indicated.
* Pregnancy or breastfeeding (pregnant or breastfeeding women are excluded from this study because oral THU-Dec has the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential, risk for adverse events in nursing infants secondary to treatment of the mother with oral THU-Dec, breastfeeding should be discontinued if the mother is treated with oral THU-Dec.
* Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
* Receiving other investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Objective Response by Revised Response Criteria for Malignant Lymphoma | Up to 52 weeks

SECONDARY OUTCOMES:
Complete Response | Up to 52 weeks
  Complete disappearance of all detectable clinical evidence of disease, and disease-related symptoms if present prior to therapy
Partial Response | Up to 52 weeks
  A > 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or extranodal masses. These nodes should be selected according to the following: (a) they should be clearly measurable in at least 2 perpendicular dimensions; (b) they should include mediastinal and retroperitoneal areas of disease whenever these sites are involved.
  No increase in the size of other nodes, liver or spleen.
  Bone marrow assessment is irrelevant for determination of a PR if the sample was positive prior to treatment. However, if positive, the cell type should be specified, e.g. large-cell lymphoma or small cleaved cell lymphoma.
  No new sites of disease
Stable Disease | Up to 52 weeks
  Failing to attain the criteria needed for a PR or CR, but not fulfilling those for progressive disease.
  For FDG-avid lymphomas: FDG-PET/CT should be positive at prior sites of disease with no new areas of involvement on the post-treatment CT or FDG-PET/CT.
  For variably FDG-avid lymphomas/FDG-avidity unknown: For patients without a pretreatment FDG-PET/CT scan or if the pre-treatment FDG-PET/CT was negative, there must be no change in the size of the previous lesions on the post-treatment CT scan.
Progressive Disease | Up to 52 weeks
  For determination of relapsed and progressive disease, lymph nodes should be considered abnormal if the long axis is more than 1.5 cm, regardless of the short axis. If a lymph node has a long axis of 1.1 to 1.5 cm, it should only be considered abnormal if the short axis is more than 1 cm. Lymph nodes < 1 x < 1 cm will not be considered as abnormal for relapse or progressive disease. Treatment decisions in patients with presumed refractory, relapsed or progressive disease should not be made solely on the basis of a single FDG-PET/CT scan without histologic confirmation.
Duration of response | Up to 52 weeks
  This is measured, only in responders, from the documented beginning of response (CR or PR) to the time of relapse.
Disease-free survival | Up to 52 weeks
  Survival is defined as the date of study entry to the date of death. Disease-free survival is measured from the time of occurrence of disease-free state (e.g. the adjuvant setting following surgery or radiation therapy) or attainment of a complete remission) to disease recurrence or death from lymphoma or acute toxicity of treatment. This definition may be complicated by deaths that occur during the follow-up period that are unrelated to the lymphoma and there is controversy as to whether such deaths should be considered as events or censored at the time of occurrence. Whereas it is often possible to identify those deaths related to the lymphoma, there is the potential for bias in the attribution of deaths.
Disease-specific survival | Up to 52 weeks
  Disease-specific survival (e.g., lymphoma-specific survival, cause-specific survival) is potentially subject to bias because the exact cause of death is not always easy to ascertain. To minimize the risk of bias, the event should be recorded as death from lymphoma, or from toxicity from the drug. Death from unknown causes should be attributed to the drug. For certain trials, time to next lymphoma treatment may be of interest, defined as time from the end of primary treatment until the initiation of the next therapy.
Progression-free survival | Up to 52 weeks
  Progression-free Survival (PFS) is defined as the time from entry onto study until lymphoma progression or death from any cause. PFS reflects tumor growth and, therefore, occurs prior to the endpoint of overall survival. In addition, PFS is not confounded by the administration of subsequent therapy. Whether a prolongation of PFS represents direct clinical benefit or a surrogate for clinical benefit depends on the magnitude of the effect and the risk-benefit ratio of the therapy under investigation. Unlike survival, the precise date of progression is generally unknown. It may be defined as the first date of documentation of a new lesion or enlargement of a previous lesion, or the date of the scheduled clinic visit immediately after radiologic assessment has been completed. Where there is missing information, censoring of the data may be defined as the last date at which progression status was adequately assessed or the first date of unscheduled new anti-lymphoma treatment.
Time to progression | Up to 52 weeks
  Time to progression (TTP) is defined as the time from study entry until lymphoma progression or death due to lymphoma. In TTP, deaths from other causes are censored either at the time of death or at an earlier time of assessment, representing a random pattern of loss from the study. TTP is not as useful as PFS unless the majority of deaths on a study are unrelated to the lymphoma due to the efficacy of the treatment and/or prolonged follow up
Time to treatment failure | Up to 52 weeks
  Time to treatment failure (event-free survival) is measured from the time from study entry to any treatment failure including discontinuation of treatment for any reason, such as disease progression, toxicity, patient preference, initiation of new treatment without documented progression, or death. This composite endpoint is generally not encouraged by regulatory agencies because it combines efficacy, toxicity and patient withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Hill, MD, PhD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States